CLINICAL TRIAL: NCT04151524
Title: Biologic Classification of Adenocarinoma of the Esophagus and Esophagogastric Junction (AEG) Using a Novel Data-driven System: Should it Replace or Compliment the Siewert Classification?
Brief Title: Classification of Adenocarcinoma of the Esophagogastric Junction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Noel Edward Donlon, Principal Investigator, St. James's Hospital, Ireland
Other Study IDs: SJH00002
Record Dates: First submitted 2019-10-23; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Oesophagus Cancer; Barrett Esophagus; Siewert Type I Adenocarcinoma of Esophagogastric Junction; Siewert Type II Adenocarcinoma of Esophagogastric Junction; Siewert Type III Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Esophageal Neoplasms; Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Siewert classification of oesophageal cancer is the standard approach in anatomically subdividing cancer of the lower oesohagus.

DETAILED DESCRIPTION:
Retrospective review of tumour biology, pathological staging and outcomes in the participants based on Siewert classification. The investigators to scrutinise this scoring system to evaluate if it is indeed appropriate.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational study
Sampling Method: Non-Probability Sample
Enrollment: 1658 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2019-12-25 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- St. James's Hospital, Dublin, IE, Ireland

IPD SHARING:
Plan to Share IPD: No